CLINICAL TRIAL: NCT01164254
Title: Feasibility Study of a Web-Based Automated Self-Administered 24-hour Dietary Recall (ASA 24) and a Physical Activity 24-Hour Recall (ACT24)
Brief Title: Feasibility Study of a Web-Based Automated Self-Administered 24-hour Dietary Recall (ASA 24) and a Physical Activity 24-hour Recall
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908152; 08-C-N152
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-11-30

CONDITIONS: Cancer
Keywords: Exposure Assessment; Web-Based Dietary Assessment; Web-Based Physical Activity Assessment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
In spite of long-standing hypothesis relating diet and physical activity to several cancers, diet and physical activity-cancer associations have been modest at best and often inconsistent in epidemiologic studies. Investigators around the world have become increasingly concerned that error in the measurement of both diet and physical activity is compromising our ability to detect these important but modest associations. Most commonly used diet and physical activity assessment methods have been based on a relatively small set of questions (e.g. 124 food items consumed or 5-10 physical activities in the past 12 months). Recent developments in computer technology provide an opportunity to use internet-based instruments to assess an individual s diet and physical activity more accurately and cost effectively.

DETAILED DESCRIPTION:
In spite of long-standing hypothesis relating diet and physical activity to several cancers, diet and physical activity-cancer associations have been modest at best and often inconsistent in epidemiologic studies. Investigators around the world have become increasingly concerned that error in the measurement of both diet and physical activity is compromising our ability to detect these important but modest associations. Most commonly used diet and physical activity assessment methods have been based on a relatively small set of questions (e.g. 124 food items consumed or 5-10 physical activities in the past 12 months). Recent developments in computer technology provide an opportunity to use internet-based instruments to assess an individual s diet and physical activity more accurately and cost effectively.

NCI has been developing two web-based instruments, an automated self-administered 24-hour dietary recall (ASA24) and a physical activity 24-hour recall (ACT24), which can be administered several times over a year. Although these two instruments have the potential to qualitatively improve exposure assessment (at relatively low cost), they need to be evaluated for feasibility before being incorporated in cohorts on a large scale. Therefore, we propose to test ASA24 and ACT24 among AARP members aged 50 years and over to evaluate technical problems, determine response rates, and estimate the range of dietary intake and physical activity. In addition, we propose to include in this feasibility study two web-based versions of conventional questionnaires (lifestyle and medical history questionnaire and diet history questionnaire) as well as two software systems needed to conduct a web-based study (the automated Study Management System and Web Survey Management System). We will initially target 15,000 AARP members, expecting that approximately 2,000 individuals will agree to participate in the study and about 1,250 participants will complete ASA24 and ACT24 twice.

These web-based instruments and accompanying system tools represent a novel approach to carrying out diet and lifestyle research. The computerized, web-based study method can be applied to any observational study, large or small, case-control or cohort, as well as randomized controlled trials. This feasibility study will provide an opportunity to assess the feasibility of constructing large web-based cohort studies and characterize potential participants.

ELIGIBILITY:
* We will recruit 5,000 subjects from the existing NIH-AARP study participants who are currently 62 to 83 years old. To include individuals who are at least 50 years old, we will expand our recruitment effort to 10,000 new AARP members who are at least 50 years old and not currently NIH-AARP study cohort members. We will target individuals residing in one of the following states: Florida; Pennsylvania; New Jersey; Louisiana; North Carolina; California; Detroit; Michigan; and Atlanta, Georgia, Nevada, Arizona, Texas, Illinois, Washington, Wisconsin, Colorado, Connecticut, Kentucky, Utah and Massachusetts (subject to change due to availability of high-quality state cancer registries). The names and addresses of new AARP members will be provided by AARP.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2008-05-28; Study Completion 2016-11-30

CONTACTS AND LOCATIONS:
Overall Officials: Charles E Matthews, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States